CLINICAL TRIAL: NCT05910671
Title: Parent-Based Physical Activity Intervention for Black Parents and Their Preschool Aged Children
Brief Title: Parent-Based Physical Activity Intervention for Black Families
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit participants due to COVID affective the target population
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Katrina DuBose, Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-001263
Record Dates: First submitted 2023-06-06; First posted 2023-06-20 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Physical Inactivity
Keywords: Physical Activity; Black; Families; Intervention
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Phone Calls and Notebook (Experimental): The intervention will last 8 weeks. As part of the intervention the participants (parents) will receive a notebook with weekly newsletters that discuss behavioral strategies for physical activity changes, note pages, listing of local parks, and age-appropriate physical activities that parents and young children can do together. The intervention group will also have individual weekly telephone meetings with a physical activity coach. The weekly meeting is expected to last approximately 30 minutes. During this meeting, participants will discuss that week's behavioral strategy to promote physical activity, report on the past week's physical activity goals, failures and successes, and set goals for the next week. Each week parents will be asked to set a goal to be physically active with their child and a goal to be physically active alone.
  Interventions: Behavioral: Physical Activity Phone Calls and Notebook
- Control (No Intervention): During the 8 weeks the participants in the control group will neither receive the intervention material nor have any contact with physical activity coaches. They will continue interacting with their young child as normal.

INTERVENTIONS:
Behavioral: Physical Activity Phone Calls and Notebook — This intervention encouraged parents to model physical activity behaviors and co-participate in physical activity with their young child. Each week behavioral strategies for promoting physical activity change will be discussed to help parents work towards meeting their activity goals. As part of the physical activity intervention parents will receive a physical activity notebook that has newsletters, suggested activities that can be done with their child, and other material that will help the parent and child be active active together. The behavioral strategies and the information in the notebook will will be discussed weekly for 30 minutes via telephone.
  Arms: Physical Activity Phone Calls and Notebook

SUMMARY:
This study is an 8-week parent-based physical activity intervention focusing on increasing physical activity in preschool-aged children. The participants will be randomized into two groups: control and intervention. During the 8 weeks those in the intervention group will receive weekly newsletters and have weekly phone calls with a physical activity coach. The material in weekly newsletters and focus of the phone calls will be on behavior changes related to physical activity. Parents will be encouraged to complete physical activity alone and with their child. The control group will not have any contact with study staff during the 8-week intervention and continue with normal behaviors. Physical activity levels in the parents and children will be measures before and after the intervention.

DETAILED DESCRIPTION:
This research will examine how preschool-aged children's physical activity levels will be affected based off an intervention that encourages physical activity engagement between parents and children. A secondary purpose is to determine if the intervention impacts the children's body mass index. Black parents with a child between the ages of 2-5 will be recruited to participate in the study. Before the intervention begins, parents will complete questionnaires on demographics, health history, physical activity knowledge, family physical activity, and parenting styles. Then both parents and children will have weight, height, resting heart rate and blood pressure measured. Finally, the parents and children will be given physical activity monitors to wear for 7 days. After wearing the activity monitors the dyads will be randomized into either a control or intervention group. The control group will continue with their normal activities for 8 weeks. Those in the intervention group will receive weekly newsletters and a 30-min/week telephone call with an activity coach over 8 weeks. The newsletters and phone calls will discuss information related to physical activity change. After the 8-week time period, all parent-child dyads will complete the same questionnaires and measurements and wear the activity monitors again.

ELIGIBILITY:
Inclusion Criteria:

* adults who are 19 years old or older
* adult has a child who is between 2-5 years old
* child must be living with the parent
* parent identifies as Black/African American

Exclusion Criteria:

* parent is currently meeting physical activity recommendations
* parent is currently pregnant or < 6 weeks post-pregnancy
* child has condition that restricts physical activity
* parent is unable to speak or write in English

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
change in parent physical activity | week 1 and week 10
  minutes spent in moderate to vigorous physical activity
change in child physical activity | week 1 and week 10
  minutes spent in total physical activity

SECONDARY OUTCOMES:
change in family physical activity | week 1 and week 10
  minutes spent in physical activity spent between parent and child

CONTACTS AND LOCATIONS:
Overall Officials: Katrina D DuBose, PhD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States